CLINICAL TRIAL: NCT05703659
Title: B2BBB: Baby 2 Baby Beneficial Bacteria
Brief Title: Baby 2 Baby Beneficial Bacteria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit a sufficient number of women in one month to start the lactation support groups.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB202200652
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Transmission
Keywords: Transmission; Beneficial bacteria; Probiotic; B. longum subsp. infantis; L. reuteri; breastfed infants

STUDY DESIGN:
Intervention Model Description: Primary Purpose of this study is epidemiological, and to determine if probiotic species can transmit between infants whose microbiomes are still developing.
  Mothers and infant dyads will be enrolled and attend 5 weekly lactation support group sessions. After the first session, infants will be randomized to receive 1 of 2 probiotics. Both probiotics are marketed in the US as dietary supplements for infants. At the first support group session and at the final session, infant fecal samples and mother's milk samples will be collected and tested for detectable levels of both probiotics to determine if horizontal transmission of the probiotic species occurred in the setting of a lactation support group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMO consuming bacteria (Experimental): Infants will given a daily HMO consuming probiotic (B. infantis) for four weeks
  Interventions: Dietary Supplement: B. longum subsp. infantis
- Non-HMO consuming bacteria (Experimental): Infants will be given a daily non-HMO consuming probiotic (L. reuteri) for four weeks
  Interventions: Dietary Supplement: L. reuteri probiotic

INTERVENTIONS:
Dietary Supplement: B. longum subsp. infantis — Infants will receive 1 dose of a B. infantis probiotic daily for 4 weeks
  Arms: HMO consuming bacteria
Dietary Supplement: L. reuteri probiotic — Infants will receive 1 dose of an L. reuteri probiotic daily for 4 weeks
  Arms: Non-HMO consuming bacteria

SUMMARY:
The investigators will recruit mother-infant dyads to attend weekly lactation support groups and randomize infants to receive either an HMO consuming or non-HMO consuming probiotic. The investigators will collect infant stool before and after support group attendance. The investigators will use qPCR and metagenomic sequencing to test if the study probiotics or other bacteria transmit between infants. The investigators anticipate HMO consuming bacteria will and non-HMO consuming bacteria will not transmit between infants.

DETAILED DESCRIPTION:
The investigators will recruit mother-infant dyads to attend weekly lactation support groups for five weeks and randomize infants to receive either an HMO consuming (B. longum subsp. infantis) or non-HMO consuming (L. reuteri) probiotic. The investigators will collect a baseline infant stool sample and maternal milk sample before attendance at the first lactation support group meeting. At the first support group meeting, mothers will be provided with the open label probiotic their infant was randomized to receive, and will give the probiotic daily for the next 28 days. The investigators will collect a second infant stool sample and a second milk sample at the final lactation support group meeting. The investigators will use qPCR and metagenomic sequencing to test if the study probiotics or other bacteria transmit from the infants who received a specific species to the infants who did not receive that species. We will also test to see if the probiotic given to infants is detectable in milk samples. The investigators anticipate HMO consuming bacteria will and non-HMO consuming bacteria will not transmit between infants.

ELIGIBILITY:
NOTE: Age limits listed are for mothers. For infants, age limits are a minimum of 1 day and a maximum of 1 month

Inclusion Criteria:

* Healthy singleton pregnancy, term delivery (>= 36 weeks corrected gestational age)
* Maternal intent to exclusively breastfeed for the first six months of infant life (intent to breastfeed for six months correlates with longer duration of breastfeeding, this increases the chance that mothers will still be breastfeeding at the end of the study)
* Maternal vaccination against COVID19 (2 doses Pfizer or Moderna and within 6 months of second dose or 2 doses Pfizer or Moderna and booster.) COVID vaccination is required for maternal participation as this is a study meant to enable transmission of beneficial bacteria species between infants, and infants are too young to be vaccinated.

Exclusion Criteria:

* Maternal drug abuse
* Infant congenital abnormalities
* Infant age greater than 1 month at first lactation support group meeting (younger infants will have less developed microbiomes, increasing the chance of successful transmission of bacteria)
* Intent to provide a non-study probiotics to the infant
* Known immunocompromised status of the infant.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Transmission of probiotics to non-supplemented infants | 4 weeks
  Percentage of infants with detectable levels of B. infantis who were not given a B. infantis probiotic and were not colonized by B. infantis at baseline OR percentage of infants with detectable levels of L. reuteri who were not given an L. reuteri probiotic and were not colonized by L. reuteri at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Taft, BA, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No